CLINICAL TRIAL: NCT06068972
Title: A Retrospective Database Analysis of the Impact of Fluorescence Imaging of Bacterial Presence, Location, and Load on Wound Healing, Antibiotic Usage, and Infection Related Complications
Brief Title: Retrospective Database Review at LTC and SNFs
Status: Completed | Type: Observational
Sponsor: Wound Care Plus, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 22-001
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Non-Healing Ulcer of Skin; Autofluorescence Imaging
Keywords: chronic wounds; bacterial loads; fluorescence imaging; MolecuLight; long-term care; skilled nursing facility
MeSH Terms: interventions — Optical Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- MolecuLight cohort: The MolecuLight bacterial imaging procedure was used in combination with standard of care clinical wound assessment.
  Interventions: Device: MolecuLight
- Standard of Care cohort: Standard of care clinical wound assessment.

INTERVENTIONS:
Device: MolecuLight — Point-of-care fluorescence imaging of high bacterial loads
  Other Names: Autofluorescence imaging
  Groups: MolecuLight cohort

SUMMARY:
The goal of this observational study is to compare the differences in wound outcomes when the MolecuLight imaging procedure is used in combination with standard of care wound assessment in long term care and skilled nursing facilities. The main outcome studied is healing of ulcers after 12-weeks, along with other outcomes such as occurrence of infection, complications, and antimicrobial use. Medical records from the past were reviewed, where patients receiving the MolecuLight procedure were compared to those who did not.

ELIGIBILITY:
Inclusion Criteria:

* Were first treated by Wound Care Plus LLC during time periods from Jan 2019-Feb 2020 (standard of care cohort) and May 2021-Mar 2022 (Moleculight cohort)
* Received at least one debridement, as indicated by CPT codes 11042, 11045, 97597, and/or 97598, during the study admission period
* Were treated by a Wound Care Plus LLC provider for at least 4 calendar weeks during the study period
* Were treated in a SNF or LTC setting during the study admission period
* Were covered by Medicare of Missouri during the study admission period
* Had at least one chronic ulcer with ICD-10 diagnosis codes L89, L97, L98, or L97/L98 in combination with E11 during the study admission period
* MolecuLight cohort ONLY: at least one MolecuLight imaging procedure during the study admission period, indicated by CPT code 0598T

Exclusion Criteria:

* Did not receive at least one debridement, as indicated by CPT codes 11042, 11045, 97597, and/or 97598, during the study admission period
* Received care from Wound Care Plus LLC for less than 4 calendar weeks during the study admission period
* Were not treated in a SNF or LTC setting during the study admission period
* Were not covered by Medicare of Missouri during the study admission period
* Did not have a chronic ulcer with ICD-10 diagnosis codes L89, L97, L98, or L97/L98 in combination with E11 during the study admission period
* MolecuLight cohort ONLY: did not receive a MolecuLight imaging procedure during the study admission period, indicated by CPT code 0598T

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Medicare beneficiaries in the state of Missouri who began receiving wound care (admission period) from Wound Care Plus LLC providers during time periods from Jan 2019-Feb 2020 (standard of care cohort) and May 2021-March 2022 (Moleculight cohort).
Sampling Method: Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Proportion of wounds healed | 12-weeks
Time to healing among wounds healed during study period | 2019-2022

SECONDARY OUTCOMES:
Occurrence of wound-related infection, infection complications, antimicrobial use over the study period | 2019-2022

CONTACTS AND LOCATIONS:
Locations (1):
- Wound Care Plus, LLC, Blue Springs, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
To protect patient confidentiality, the study data are not publicly available; however they are available from the authors upon reasonable request and with permission of Wound Care Plus, LLC.